CLINICAL TRIAL: NCT00242762
Title: A Phase II Study to Evaluate the Safety and Efficacy of the Combination of ZD1839 (IRESSA™), Docetaxel and Cisplatin in Subjects With Recurrent and/or Metastatic Head and Neck Cancer
Brief Title: ZD1839 (IRESSA™) in Combination With Docetaxel & Cisplatin in Subjects With Metastatic Head & Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0504
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Neoplasms; Cancer of Head and Neck; Head and Neck Cancer; Head Cancer; Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Gefitinib; Docetaxel; Cisplatin

INTERVENTIONS:
Drug: ZD1839 (IRESSA™)
Drug: Docetaxel
Drug: Cisplatin

SUMMARY:
The primary objective of the study is to evaluate the activity of the combination ZD1839, docetaxel and cisplatin in subjects with recurrent and/or metastatic head and neck cancer by estimating the objective response rate (complete response [CR] and partial response [PR]) at study closure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 and 70 years, inclusive
2. Histologically- or cytologically-confirmed recurrent and/or metastatic SCCHN
3. Primary tumour site of oral cavity, oropharynx, hypopharynx or larynx
4. At least one uni-dimensionally measurable lesion according to the RECIST
5. World Health Organisation (WHO) performance status (PS) of 0 or 1
6. No previous chemotherapy for recurrent or metastatic disease
7. Before subject registration a quality of life questionnaire should be completed

Exclusion Criteria:

1. Previous chemotherapy for recurrent or metastatic disease
2. Less than 6 months since prior induction or adjuvant platinum and/or taxanes chemotherapy
3. Known severe hypersensitivity to ZD1839 or any of the excipients of this product
4. Known, severe hypersensitivity to docetaxel or cisplatin or any of the excipients of these products, or to other drugs formulated with polysorbate 80
5. Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
6. Any unresolved chronic toxicity greater than common toxicity criteria (CTC) grade 2 from previous anticancer therapy (except alopecia)
7. Absolute neutrophil count (ANC) less than 1.5 x109/litre (L), platelets less than 100 x 109/L or haemoglobin less than 10 g/dl
8. Serum bilirubin greater than the upper limit of the reference range (ULRR)
9. Serum creatinine greater than 1.5 mg/dl despite adequate rehydration
10. Creatinine clearance less than 60 ml/min assessed in over a 24 hour urine collection
11. As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease)
12. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 1.5 times the ULRR or alkaline phosphatase (ALP) greater than 2.5 times the ULRR
13. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study
14. Pregnancy or breast feeding (women of child-bearing potential)
15. Concomitant use of phenytoin, carbamazepine, rifampicin, or barbiturates, or St John's Wort
16. Treatment with a non-approved or investigational drug within 30 days before Day 1 of study treatment
17. Any evidence of clinically active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic need not be excluded

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Objective tumour response (CR and PR) at study closure based on the Response Evaluation Criteria in Solid Tumours (RECIST)

SECONDARY OUTCOMES:
PFS
Overall survival
Incidence of DLT during the first cycle of study treatment
Nature, incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Spain Medical Director, MD, Study Director — AstraZeneca
Locations (4):
- Spain (4):
  - Research Facility, Granada
  - Research Facility, Madrid
  - Research Facility, Murcia
  - Research Site, Seville